CLINICAL TRIAL: NCT05797896
Title: A Multicentre, Natural History, Non-interventional Study Evaluating Biomarkers In Participants With Geographic Atrophy(GA) Secondary To Age-Related Macular Degeneration (AMD)
Brief Title: Investigating Geographic Atrophy Insights (i-GAIN) Natural History Study
Acronym: i-GAIN
Status: Active, not recruiting | Type: Observational
Sponsor: Complement Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: IGS01; i-GAIN (Other: Complement Thearapeutics)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Dry Age-related Macular Degeneration; Geographic Atrophy; Retinal Disease; Macular Degeneration; Macular Atrophy; Retinal Degeneration; Eye Diseases
Keywords: Dry Age-related Macular Degeneration; Geographic Atrophy; Retinal Disease; Macular Degeneration; Macular Atrophy; Retinal Degeneration; Eye Diseases; AMD; GA
MeSH Terms: conditions — Geographic Atrophy; Retinal Diseases; Macular Degeneration; Anetoderma; Retinal Degeneration; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An observational study to investigate the natural history and evaluate biomarkers of participants with geographic atrophy secondary to age-related macular degeneration

DETAILED DESCRIPTION:
Prospective, observational study to assess the relationships between circulating levels of complement proteins measured using the Complement Precision Medicine (CPM) Platform, genetic profile and lesion progression in subjects with Geographic Atrophy (GA) secondary to Age-related Macular Degeneration (AMD) up to a 24-month period

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of bilateral GA due to AMD as confirmed by fundoscopy and imaging at Screening
2. GA lesion sizes of ≥ 1.25 mm2 to ≤ 17 mm2 (approximately 1-7 disc diameters) in at least one eye as per Central Reading Center
3. Willing and able to provide written informed consent
4. Male or female aged 65 years and over

Exclusion Criteria:

1. History of neovascular (wet) AMD or presence of neovascular (wet) AMD in either eye confirmed by fundoscopy at screening and/or any pre-existing retinal imaging
2. History of intravitreal (IVT) injection in the study eye. Note: Intravitreal treatment with pegcetacoplan (Syfovre®) and avacincaptad pegol (IzervayTM) if approved within the participant's country of origin AND if deemed necessary by the Principal Investigator (PI) is allowed in the fellow eye only. IVT injections in the study eye are prohibited.
3. History of uveitis or endophthalmitis
4. High myopia (more than 6 diopter) in the study eye
5. Any ocular pathology which would impede clear imaging of the macula, e.g. intra-ocular opacities
6. Macular changes from causes other than AMD
7. Diabetic retinopathy in either eye. Note: Presence of systemic diabetes with no retinopathy is not exclusionary
8. Any other physical condition which would prevent the participant from undertaking imaging procedures
9. Any cell or gene therapy in either eye

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Approximately 250 participants, age 65 years and older, with bilateral GA due to AMD will be accrued.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Levels of complement proteins | Month 6, 12,18, 24
  To assess the correlation between circulating levels of complement proteins measured using the Complement Precision Medicine (CPM) Platform and Geographic Atrophy (GA) secondary to Age-related Macular Degeneration (AMD)

SECONDARY OUTCOMES:
Geographic Atrophy | Up to 24 months
  To investigate whether there is a relationship between progression of GA and complement profile measured using the CPM platform
Genetics | Up to 24 months
  To investigate the relationship between variants in genes or loci associated with AMD and the complement profile measured using the CPM platform
Complement Proteins Intra-individual Variation | Up to 24 months
  To determine the intra-individual variation in complement profile using the Complement Precision Medicine (CPM) Platform, in participants with GA
Complement Proteins and Progression of GA | Up to 24 months
  To investigate whether there is a relationship between progression of GA and complement profile measured using the Complement Precision Medicine (CPM) platform
Choroidal Blood Flow and Genetics | Up to 24 months
  To investigate the relationship in genes or loci associated with AMD and choroidal blood flow and structure
Choroidal Blood Flow and GA Lesion Progression | Up to 24 months
  To investigate the relationships between choroidal blood flow and structure and GA lesion progression
CRP Levels | Up to 24 months
  To observe the influence of any past or concurrent illnesses, in particular inflammation-related illnesses, rise in serum CRP or of any medications on complement profile using the CPM Platform

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ugarte, Principal Investigator — Manchester Royal Eye Hospital
Locations (22):
- United States (10):
  - Global Research Management, Glendale, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Midwest Eye Institute, Carmel, Indiana
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Sierra Eye Associates, Reno, Nevada
  - Verum Research LLC, Eugene, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Plano, Texas
  - San Antonio Eye Center, San Antonio, Texas
- United Kingdom (12):
  - Belfast City Hospital, Belfast
  - Bradford Royal Infirmary, Bradford
  - Frimley Park Hospital, Frimley
  - Gloucestershire Royal Hospital, Gloucester
  - Liverpool Hospital, Liverpool
  - Moorfields Eye Hospital, London
  - Western Eye Hospital, London
  - Manchester Royal Eye Hospital, Manchester
  - Newcastle Hospital, Newcastle
  - Nottingham City Hospital, Nottingham
  - University Hospital Southampton, Southampton
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: No